CLINICAL TRIAL: NCT01977469
Title: Impact of Aerobic and High and Low Resistance Training on Daily Life Activities and BODE Index COPD Patients
Brief Title: Randomized Controlled Study to Investigate the Impact of Different Intensities Training on ADL and BODE Index in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Valeria Amorim Pires Di Lorenzo, PhD, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EditalUniversal2011
Record Dates: First submitted 2013-09-20; First posted 2013-11-06 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Activities of Daily Living; Mortality; Strength Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low intensity resistance training (Experimental): Low intensity resistance training + aerobic training
  Interventions: Behavioral: Low intensity resistance training; Behavioral: Aerobic training
- High intensity resistance training (Experimental): High intensity resistance training + aerobic training
  Interventions: Behavioral: High intensity resistance training; Behavioral: Aerobic training

INTERVENTIONS:
Behavioral: Low intensity resistance training — The LIRT group initiated the resistance training for UL with 30% of the 1RM, with 5% increases each nine sessions; therefore, the maximum load was 45% of the 1RM. The LL training initiated with 30% of the 1RM, increasing 7% each nine sessions, thus, the maximum load was 51% of the 1RM. Each exercise session consisted of three sets of 15 repetitions, with a 2 minutes interval between sets.
  Other Names: LIRT; Low-intensity resistance training
  Arms: Low intensity resistance training
Behavioral: High intensity resistance training — the initial load for HIRT group was 60% of 1RM for UL with 5% increases each nine sessions; therefore, the maximum load reached 75% of the 1RM. The LL training initiated with 60% of the 1RM with 7% increments each nine sessions, as a result, the maximum load after 36 sessions was 81% of the 1RM. These patients underwent three sets of eight repetitions, with two minutes intervals between sets.
  Other Names: HIRT; High-intensity resistance training
  Arms: High intensity resistance training
Behavioral: Aerobic training — Patients underwent an aerobic training in cycle ergometer, with load intensity determined as the same load the patient presented a VO2 value of 70-80% of the peak VO2 obtained in the symptom-limited CPET. Each session of aerobic training lasted 20-30min according to patient's tolerance.
  Other Names: AT

SUMMARY:
The local and systemic manifestations that affect patients with Chronic Obstructive Pulmonary Disease (COPD) cause severe dyspnoea and limitation of functional capacity, leading to impairment in the performance of activities of daily living (ADL). The combination of aerobic and resistance training, for both upper limbs (UL) and lower limbs (LL), appears to be the physiologically most complete resource for improving quality of life and increased survival of these patients. Therefore, the aim of the study is to assess the impact of aerobic and resistance training of different intensities on the performance and dyspnoea during activities of daily living and prediction of mortality in patients with COPD. There will be include 45 COPD patients with moderate to severe obstruction, aged between 50-80 years of both gender. All patients will undergo to the following assessments and reassessments: history and anthropometric data, Scale London Chest Activity of Daily Living Scale (LCADL), modified Medical Research Council (mMRC), BODE index, test peripheral muscle strength, mobility and balance tests, 6-minute walk test (6MWT), Circuit ADL Test, 1 repetition maximum (1RM) and Incremental Cardiopulmonary Testing (ICPT). Patients will be randomly divided into two groups and undergo to the treatment program will consist of sessions lasting approximately 1 hour, three times a week for 12 consecutive weeks, totaling 36 sessions. All patients will undergo general stretching and aerobic training on a cycle ergometer with the intensity between 70-80 % of the maximum load achieved in ICPT. After aerobic training, a group of patients will achieve a protocol of low-intensity resistance training (LI-RT), with emphasis on gaining muscle strength, and the other group will be submitted to a protocol of high intensity (HI-RT), aiming greater gain in muscle strength. The calculation of the intensity of training will be conducted by the 1RM test. After the training protocol, it is expected to find improved performance and dyspnoea during activities of daily living and reduction of BODE index for both groups, however, it is expected that the group of low-intensity resistance training presents greater benefits in ADL.

ELIGIBILITY:
Inclusion Criteria:Patients both genders, with a clinical diagnosis of COPD confirmed by post bronchodilator spirometry administered by a pneumologist, classified as moderate to very severe obstruction in accordance with the GOLD criteria; ex- or non-smokers; oxygen dependent or not; clinically stable; no history of infection and no exacerbation of respiratory symptoms or changes in medication for at least two months before the study and that no present cardiac, rheumatic or an associated orthopedic disease that prevent them from performing the proposed evaluation tasks.

Exclusion Criteria:Patients who present respiratory, cardiac, rheumatic, musculoskeletal, orthopedic and neuromuscular sequels that may prevent the testing and intervention proposal; that to modify the type of medication during the study; in cases of uncontrolled hypertension or refusal to provide consent proposed in the Resolution of National Council of Health.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Saturation During Activities of Daily Living | Baseline and after 36 sessions, an average of 3 months
  TThe ADL performance was assessed by an adapted laboratory circuit of ADL, including: Showering, lifting and lowering containers on a shelf above the shoulder girdle, and raising and lowering pots on a shelf below the pelvic girdle.
  Oxygen saturation (SpO2, %) was assessed by pulse oxymeter.
Change in Ventilation During Activities of Daily Living | Baseline and after 36 sessions, an average of 3 months
  The ADL performance was assessed by an adapted laboratory circuit of ADL, including: Showering, lifting and lowering containers on a shelf above the shoulder girdle, and raising and lowering pots on a shelf below the pelvic girdle.
  Ventilation (VE-l/min) was captured by a portable metabolic system.
Change in Oxygen Consumption During Activities of Daily Living | Baseline and after 36 sessions, an average of 3 months
  The ADL performance was assessed by an adapted laboratory circuit of ADL, including: Showering, lifting and lowering containers on a shelf above the shoulder girdle, and raising and lowering pots on a shelf below the pelvic girdle. Gas exchange (oxygen consumption - VO2-l/min) was captured by a portable metabolic system.
Change in Dyspnea Related During Activities of Daily Living | Baseline and after 36 sessions, an average of 3 months
  Dyspnea in ADL was assessed by London Chest Activity of Daily Living Scale(LCADL), that consists 15 quantitative questions of 4 domains: self-care, domestic, physical, and leisure. Subjects indicate a score of 0-5, in a total of 75 points. A higher total score indicates greater limitation in performing ADL due to dyspnea.

SECONDARY OUTCOMES:
Change in BODE index | Baseline and after 36 sessions, an average of 3 months
  In order to calculate the BODE index, the following variables were considered: BMI (body mass index), forced expiratory volume in one second, as the percentage of the predicted value (pred FEV1 %), mMRC score (modified Medical Research Council Scale) and in the 6MWD (Six-Minute Walk Distance). The score was considered according to the results obtained from the four variables (0-3 for FEV1; 0-3 for mMRC; 0-3 for 6MWD and 0-1 for BMI), and total score ranged from 0 to 10 (higher scores indicate more severity).

CONTACTS AND LOCATIONS:
Overall Officials: Valéria Amorim Pires Di Lorenzo, PhD, Study Director — Universidade Federal de Sao Carlos; Júlia Gianjoppe dos Santos, PhD, Principal Investigator — Universidade Federal de Sao Carlos; Marina Sallum Barusso, MsC, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Special Respiratory Physiotherapy Unit of the Federal University of São Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Beauchamp MK, O'Hoski S, Goldstein RS, Brooks D. Effect of pulmonary rehabilitation on balance in persons with chronic obstructive pulmonary disease. Arch Phys Med Rehabil. 2010 Sep;91(9):1460-5. doi: 10.1016/j.apmr.2010.06.021. PMID 20801268
- [Background] Bernard S, LeBlanc P, Whittom F, Carrier G, Jobin J, Belleau R, Maltais F. Peripheral muscle weakness in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1998 Aug;158(2):629-34. doi: 10.1164/ajrccm.158.2.9711023. PMID 9700144
- [Background] Clini E, Costi S, Romagnoli M, Florini F. Rehabilitation of COPD patients: which training modality. Monaldi Arch Chest Dis. 2004 Jul-Sep;61(3):167-73. doi: 10.4081/monaldi.2004.697. PMID 15679011
- [Background] Garrod R, Bestall JC, Paul EA, Wedzicha JA, Jones PW. Development and validation of a standardized measure of activity of daily living in patients with severe COPD: the London Chest Activity of Daily Living scale (LCADL). Respir Med. 2000 Jun;94(6):589-96. doi: 10.1053/rmed.2000.0786. PMID 10921765
- [Background] Eisner MD, Blanc PD, Yelin EH, Sidney S, Katz PP, Ackerson L, Lathon P, Tolstykh I, Omachi T, Byl N, Iribarren C. COPD as a systemic disease: impact on physical functional limitations. Am J Med. 2008 Sep;121(9):789-96. doi: 10.1016/j.amjmed.2008.04.030. PMID 18724969
- [Background] Man WD, Kemp P, Moxham J, Polkey MI. Skeletal muscle dysfunction in COPD: clinical and laboratory observations. Clin Sci (Lond). 2009 Aug 17;117(7):251-64. doi: 10.1042/CS20080659. PMID 19681758
- [Background] Ortega F, Toral J, Cejudo P, Villagomez R, Sanchez H, Castillo J, Montemayor T. Comparison of effects of strength and endurance training in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2002 Sep 1;166(5):669-74. doi: 10.1164/rccm.2107081. PMID 12204863
- [Background] O'Shea SD, Taylor NF, Paratz JD. Measuring muscle strength for people with chronic obstructive pulmonary disease: retest reliability of hand-held dynamometry. Arch Phys Med Rehabil. 2007 Jan;88(1):32-6. doi: 10.1016/j.apmr.2006.10.002. PMID 17207672
- [Background] Panton LB, Golden J, Broeder CE, Browder KD, Cestaro-Seifer DJ, Seifer FD. The effects of resistance training on functional outcomes in patients with chronic obstructive pulmonary disease. Eur J Appl Physiol. 2004 Apr;91(4):443-9. doi: 10.1007/s00421-003-1008-y. Epub 2003 Nov 25. PMID 14639479
- [Background] Rabe KF, Hurd S, Anzueto A, Barnes PJ, Buist SA, Calverley P, Fukuchi Y, Jenkins C, Rodriguez-Roisin R, van Weel C, Zielinski J; Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2007 Sep 15;176(6):532-55. doi: 10.1164/rccm.200703-456SO. Epub 2007 May 16. PMID 17507545
- [Background] Swallow EB, Reyes D, Hopkinson NS, Man WD, Porcher R, Cetti EJ, Moore AJ, Moxham J, Polkey MI. Quadriceps strength predicts mortality in patients with moderate to severe chronic obstructive pulmonary disease. Thorax. 2007 Feb;62(2):115-20. doi: 10.1136/thx.2006.062026. Epub 2006 Nov 7. PMID 17090575
- [Background] Troosters T, Casaburi R, Gosselink R, Decramer M. Pulmonary rehabilitation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2005 Jul 1;172(1):19-38. doi: 10.1164/rccm.200408-1109SO. Epub 2005 Mar 18. No abstract available. PMID 15778487
- [Background] Velloso M, Stella SG, Cendon S, Silva AC, Jardim JR. Metabolic and ventilatory parameters of four activities of daily living accomplished with arms in COPD patients. Chest. 2003 Apr;123(4):1047-53. doi: 10.1378/chest.123.4.1047. PMID 12684292
- [Background] Wedzicha JA, Bestall JC, Garrod R, Garnham R, Paul EA, Jones PW. Randomized controlled trial of pulmonary rehabilitation in severe chronic obstructive pulmonary disease patients, stratified with the MRC dyspnoea scale. Eur Respir J. 1998 Aug;12(2):363-9. doi: 10.1183/09031936.98.12020363. PMID 9727786
- [Derived] Barusso MS, Gianjoppe-Santos J, Basso-Vanelli RP, Regueiro EM, Panin JC, Di Lorenzo VA. Limitation of Activities of Daily Living and Quality of Life Based on COPD Combined Classification. Respir Care. 2015 Mar;60(3):388-98. doi: 10.4187/respcare.03202. Epub 2014 Dec 9. PMID 25492955